CLINICAL TRIAL: NCT05676489
Title: MeFAMP for Imaging System A Amino Acid Transport in Primary and Metastatic Brain Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R22-225
Record Dates: First submitted 2022-12-12; First posted 2023-01-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers; Recurrent Glioma; Brain Metastases From Extra-cranial Solid Tumors
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Volunteers (cohort 1) (Experimental): Whole Body Dosimetry for healthy volunteers
  Interventions: Drug: [F-18]MeFAMP PET
- High Grade Glioma (cohort 2) (Experimental): Recurrent high grade glioma after radiation therapy
  Interventions: Drug: [F-18]MeFAMP PET
- Brain Metastasis (cohort 3) (Experimental): Brain metastases from extra-cranial solid tumors before and after radiation therapy
  Interventions: Drug: [F-18]MeFAMP PET

INTERVENTIONS:
Drug: [F-18]MeFAMP PET — Study participants will receive the fluorine-18 labeled system A amino acid transport substrate, (R)-3-[F-18]fluoro-2-methyl-2-(methylamino)propanoic acid ([F-18]MeFAMP), for positron emission tomography (PET). Participants in Cohorts 1 and 2 will receive a single administration of the study drug. Participants in cohort 3 will receive 2 administrations of the study drug, once before standard of care radiation therapy for brain metastases and once after.

SUMMARY:
This first-in-human study will establish the human safety and radiation dosimetry of the system A amino acid transport substrate, (R)-3-[F-18]fluoro-2-methyl-2-(methylamino)propanoic acid ([F-18]MeFAMP), for positron emission tomography (PET) imaging of primary and metastatic brain tumors. This study will include 3 cohorts: healthy volunteers for whole body dosimetry estimates (n=6-8, Dosimetry Cohort), patients undergoing evaluation for recurrent high grade glioma after radiation therapy (n=10, high grade glioma (HGG) Cohort), and patients with brain metastases from extra-cranial solid tumors before and after radiation therapy (n=10, Metastasis Cohort). Exploratory assessment of the diagnostic accuracy of MeFAMP for distinguishing recurrent/progressive brain tumors from radiation-related treatment effects will also be performed for subsequent trial design. The study will complete accrual and safety assessment in the Dosimetry Cohort before recruiting for the HGG and Metastasis Cohorts.

ELIGIBILITY:
Inclusion Criteria for all cohorts:

1. 18 years of age or older at the time of enrollment
2. Females with childbearing potential must have a negative urine human chorionic gonadotropin (hCG) test on the day of procedure or a serum hCG test within 48 hours prior to the administration MeFAMP.
3. Must have a life expectancy greater than 12 weeks.

Exclusion Criteria for all cohorts:

1. Use of an investigational drug for any indication within 3 months prior to the imaging study.
2. Pregnancy or breast feeding
3. Inability to complete the PET scans.
4. Significant renal or hepatic dysfunction (estimated glomerular filtration rate (GFR) < 60 mL/min)
5. Any condition which may interfere with ability to participate in or complete all study-related activities as assessed by the study team.

6.4.9.3. Inclusion criteria specific to Dosimetry Cohort

1. Normal complete metabolic profile (CMP) and cell blood count (CBC) with differential at baseline.
2. Normal ECG at baseline.

Exclusion criteria specific to Dosimetry Cohort

1) Major medical problems (e.g. renal, hepatic, inflammatory) that could interfere with biodistribution of MeFAMP as assessed by the study team.

Inclusion Criteria specific to HGG Cohort

1. Grade III or Grade IV glioma previously treated with radiation therapy
2. Standard of care contrast-enhanced MRI showing an enhancing lesion at least 1-cm in maximum dimension that is equivocal or suspicious for recurrent glioma.
3. Eastern Cooperative Oncology Group (ECOG) performance score of 2 or better

Inclusion Criteria specific to Metastasis Cohort

1. At least one brain metastasis from melanoma, lung cancer (small or non-small cell), or breast cancer measuring at least 1-cm in maximum dimension on contrast-enhanced MRI
2. Plan for stereotactic radiation therapy within 2 weeks of initial MeFAMP-PET/MRI scan.
3. ECOG performance score of 2 or better

Inclusion of Women and Minorities

Patients 18 years of age or older will be eligible for study participation. No other discriminatory factors, including age, sex, or ethnic background will be used to determine eligibility. Every effort will be made to ensure that minorities are recruited for study participation.

Ages: 18 Months to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Human dosimetry for [F-18]MeFAMP. | From injection to 45 minutes, 2 hours, and 4 hours after PET agent administration.
  The changing concentrations of radioactivity in normal organs and tissues will be measured in each participant at 3 time points after [F-18]MeFAMP injection in Cohort 1. These data will be used to estimate human dosimetry as effective dose in milliSieverts.
Safety of [F-18]MeFAMP | Lab values, ECG and adverse events will be assessed on the day of the study before and after administration of [F-18]MeFAMP for cohort 1.
  Laboratory values including complete metabolic panel (CMP) and complete blood count with differential (CBC with diff) and adverse events will be assessed before and after [F-18]MeFAMP administration in cohort 1. Electrocardiograms (ECG) will also be performed before and after study drug administration in cohort 1 to assess for QT prolongation and changes in heart rate, rhythm, and ECG waveforms that could represent a safety signal due to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No